CLINICAL TRIAL: NCT01321762
Title: Effect of Pregnancy and Childbirth on the Pelvic Floor
Brief Title: Prolapse and Pregnancy Assessment
Acronym: PAPA
Status: Completed | Type: Observational
Sponsor: Croydon University Hospital (Other)
Responsible Party: Principal Investigator, Ranee Thakar, Consultant, Croydon University Hospital
Other Study IDs: 05/Q0806/9
Record Dates: First submitted 2011-03-11; First posted 2011-03-24 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Prolapse; Childbirth; Pregnancy
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Pregnant Women with singleton pregnancy

SUMMARY:
Pelvic organ prolapse (POP) is one of the most common indications for gynaecological surgery. In 1997, more than 225000 inpatient surgical procedures for POP were undertaken in USA (22.7 per 10000 women) at an estimated cost of more than one billion dollars. In the UK, the disorder accounts for 20% of the women on the waiting list for major gynaecological surgery. Vaginal birth, advancing age and increasing body mass are the most consistent risk factors. Furthermore a racial and congenital predisposition has been reported. The cause of this disorder is likely to be multifactorial and attributable to a combination of factors, varying from patient to patient.

Controversy exists as to whether the pregnancy per se rather than the mode of delivery alters the risk of POP. Caesarean section appears to protect against the development of prolapse. However, when a caesarean section is undertaken during the active stage of labour it may not be completely protective. Ideally prospective longitudinal studies are needed to study the impact of pregnancy and childbirth on pelvic organ prolapse. Unfortunately, studies to date, are small with poor follow-up and have only assessed objective outcome rendering it difficult to draw conclusions. The primary objective of our study was to objectively assess the impact of pregnancy and childbirth on pelvic organ support using the Pelvic Organ Prolapse Quantification (POPQ)System.

ELIGIBILITY:
Inclusion Criteria:

* Singleton Pregnancy

Exclusion Criteria:

* Multiple pregnancies
* Previous prolapse surgery
* Medical disorders including diabetes mellitus
* Inflammatory bowel disease
* Collagen disorders

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with uncomplicated singleton pregnancy attending the ultrasound scan clinic in the second trimester were invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2005-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Objective assessment of Prolapse using Pelvic organ prolapse Quantification System | 2nd trimester, 3rd trimester, 14 weeks, 12 months and 5 years after childbirth
  Prospective evaluation of the impact of mode of delivery on pelvic organ support using the International Continence Society recommended Pelvic Organ Prolapse Quantification system (POPQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Croydon University Hospital, Croydon, Surrey, United Kingdom